CLINICAL TRIAL: NCT00739999
Title: A 8-Week, Open-Label, Phase 1 Study To Evaluate Pharmacokinetics, Pharmacodynamics, Safety And Tolerability Of Atorvastatin In Children And Adolescents With Heterozygous Familial Hypercholesterolemia
Brief Title: 8-Week PK/PD Atorvastatin Study In Children And Adolescents With Heterozygous Familial Hypercholesterolemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: A2581172
Record Dates: First submitted 2008-08-21; First posted 2008-08-22 (Estimated); Results first posted 2010-08-20 (Estimated); Last update posted 2021-03-15 (Actual); Status verified 2021-02

CONDITIONS: Pediatric Heterozygous Hypercholesterolemia
Keywords: heterozygous familial hypercholesterolemia (HeFH); atorvastatin; pediatric
MeSH Terms: interventions — Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Other): 6-10 years will be administered with atorvastatin tablet formulation with initial doses based on age cohort.
  Interventions: Drug: Atorvastatin
- 2 (Other): 10-17 years will be administered 10-mg daily dose of atorvastatin tablet formulation.
  Interventions: Drug: Atorvastatin

INTERVENTIONS:
Drug: Atorvastatin — 6-10 years Tanner Stage 1 will be administered 5-mg daily dose of an atorvastatin pediatric tablet formulation. Dose may be doubled if subjects have not attained target LDL (<3.35 mmol/L) after 4-week treatment.
  Arms: 1
Drug: Atorvastatin — 10-17 years Tanner Stage 2 will be administered 10-mg daily dose of atorvastatin tablet formulation. Dose may be doubled if subjects have not attained target LDL (<3.35 mmol/L) after 4-week treatment.
  Arms: 2

SUMMARY:
To evaluate pharmacokinetics, pharmacodynamics, safety and tolerability of atorvastatin in children and adolescents with heterozygous familial hypercholesterolemia

ELIGIBILITY:
Inclusion Criteria:

* Genetically confirmed heterozygous familial hypercholesterolemia (HeFH) with LDL greater or equal 4 mmol/L at baseline

Exclusion Criteria:

* Evidence or history of clinically significant diseases, homozygous familial hypercholesterolemia (FH)

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 39 (Actual)
Dates: Start 2008-12; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (3):
- Pfizer Investigational Site, Québec, Quebec, Canada
- Pfizer Investigational Site, Athens, Greece
- Pfizer Investigational Site, Oslo, Norway

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A2581172&StudyName=8-Week%20PK/PD%20Atorvastatin%20Study%20In%20Children%20And%20Adolescents%20With%20Heterozygous%20Familial%20Hypercholesterolemia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled at 3 medical centers and participated in the study between 02 December 2008 and 13 May 2009.
Pre-assignment Details: Forty-five subjects were screened, and 39 subjects were assigned to study treatment.
Groups:
- Atorvastatin (5 mg, 10 mg): Tanner Stage 1: Age 6 - 10 years, at Tanner Stage 1. Initial dose 5 mg/day through Week 4; after Week 4 dose may have been doubled to 10 mg/day if target low-density lipoprotein cholesterol (LDL-C) was not attained.
- Atorvastatin (10 mg, 20 mg): Tanner Stage 2+: Age 10 - 17 years, at Tanner Stage 2+. Initial dose 10 mg/day through Week 4; after Week 4 dose may have been doubled to 20 mg/day if target LDL-C was not attained.
Period: Overall Study
Arm/Group | Atorvastatin (5 mg, 10 mg): Tanner Stage 1 | Atorvastatin (10 mg, 20 mg): Tanner Stage 2+
Started | 15 | 24
Completed | 15 | 24
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Atorvastatin (5 mg, 10 mg): Tanner Stage 1: Initial dose 5 mg/day through Week 4; after Week 4 dose may have been doubled to 10 mg/day if target LDL-C was not attained and study drug was well tolerated.
- Atorvastatin (10 mg, 20 mg): Tanner Stage 2+: Initial dose 10 mg/day through Week 4; after Week 4 dose may have been doubled to 20 mg/day if target LDL-C was not attained and study drug was well tolerated.
- Total: Total of all reporting groups
Arm/Group | Atorvastatin (5 mg, 10 mg): Tanner Stage 1 | Atorvastatin (10 mg, 20 mg): Tanner Stage 2+ | Total
Number analyzed (Participants) | 15 | 24 | 39
Age, Customized [Number; unit: participants]
  6-8 years | 7 | 0 | 7
  9-10 years | 6 | 3 | 9
  11-14 years | 2 | 14 | 16
  15-17 years | 0 | 7 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 12 | 19
  Male | 8 | 12 | 20

OUTCOME MEASURES:

1. Primary Outcome: Parent-metabolite Population Pharmacokinetic (PK) Model for Atorvastatin and Its Metabolites: Atorvastatin Apparent Clearance (CL/F)
Description: Parent-metabolite population PK model built using sparse blood samples from both Tanner Stage 1 and Tanner Stage 2+. Blood sampling times: Weeks 2 and 6: single sample between 4 and 12 hours postdose; Weeks 4 and 8: predose, 1 hour, and 2 hours postdose. Plasma samples were analyzed for atorvastatin and active hydroxyacid metabolite (o-hydroxyatorvastatin) concentrations using a validated, sensitive, and specific high-performance liquid chromatography tandem mass spectrometric method. Data presented are the result of the model used.
Time Frame: Week 2, Week 4, Week 6, Week 8
Population: Pharmacokinetic (PK) concentration population: all enrolled and treated subjects who had ≥ 1 PK concentration assessed. Active hydroxyacid metabolite p-hydroxyatorvastatin was not included in the model as originally planned as > 80% of samples were below detectable level at the doses used in this trial.
Measure: Number; unit: L/hr
Arm/Group | Atorvastatin (5 mg, 10 mg): Tanner Stage 1 | Atorvastatin (10 mg, 20 mg): Tanner Stage 2+
Number analyzed (Participants) | 15 | 24
L/hr | 553 | 543
Statistical Analysis 1: Comparison: Atorvastatin (5 mg, 10 mg): Tanner Stage 1 vs Atorvastatin (10 mg, 20 mg): Tanner Stage 2+; Atorvastatin apparent clearance (CL/F) was described as a function of body weight using an allometric equation. The estimated parameter given is an extrapolation of the model for participants who weigh 70 kg; Test type: Superiority or Other; non-linear mixed-effects model; Measures of parameter estimation uncertainty (95% CI) were determined by non-parametric bootstrap analysis; Atorvastatin CL/F based on 70 kg BW = 699, 95% CI 2-sided [570 to 881]

2. Secondary Outcome: Absolute Change From Baseline in Pharmacodynamic Responses of Low-density Lipoprotein Cholesterol (LDL-C)
Description: Low-density lipoprotein cholesterol (LDL-C) measured in millimoles per liter (mmol/L); assessments were performed in the fasting state (minimum 10-hour fast [optional at Weeks 2 and 6]). Change from baseline = value at observation minus baseline value.
Time Frame: Baseline, Week 2, Week 4, Week 6, Week 8
Population: Pharmacodynamic (PD) analysis population: all enrolled subjects who received ≥ 1 dose of study drug and had ≥ 1 PD parameter measurement.
Measure: Mean (Standard Deviation); unit: mmol/L
Groups:
- Stayed at 5 mg: Tanner Stage 1: Atorvastatin 5 mg/day
- Titrated to 10 mg: Tanner Stage 1: Atorvastatin: initial dose 5 mg/day through Week 4; after Week 4 dose was doubled to 10 mg/day if target LDL-C was not attained and study drug was well tolerated.
- Stayed at 10 mg: Tanner Stage 2+: Atorvastatin 10 mg/day
- Titrated to 20 mg: Tanner Stage 2+: Atorvastatin: initial dose 10 mg/day through Week 4; after Week 4 dose was doubled to 20 mg/day if target LDL-C was not attained and study drug was well tolerated.
Arm/Group | Stayed at 5 mg: Tanner Stage 1 | Titrated to 10 mg: Tanner Stage 1 | Stayed at 10 mg: Tanner Stage 2+ | Titrated to 20 mg: Tanner Stage 2+
Number analyzed (Participants) | 5 | 10 | 9 | 15
mmol/L
  Baseline | 4.87 (0.48) | 6.37 (1.10) | 5.11 (0.65) | 6.23 (1.00)
  Week 2 | -1.75 (0.72) | -1.62 (0.46) | -1.95 (0.52) | -1.90 (0.72)
  Week 4 | -2.07 (0.50) | -1.94 (0.56) | -2.24 (0.57) | -2.27 (1.04)
  Week 6 | -1.89 (0.42) | -2.57 (0.70) | -2.12 (0.74) | -2.55 (1.02)
  Week 8 | -1.80 (0.63) | -2.71 (0.60) | -1.99 (0.58) | -2.60 (1.01)

3. Secondary Outcome: Percent Change From Baseline in Pharmacodynamic Responses of Low-density Lipoprotein Cholesterol (LDL-C)
Description: Low-density Lipoprotein Cholesterol (LDL-C): percent (%) change from baseline by treatment over time = [LDL-C at observation minus LDL-C at Week 0] divided by LDL-C at Week 0 * 100. Assessments were performed in the fasting state (minimum 10-hour fast [optional at Weeks 2 and 6]).
Time Frame: Baseline, Week 2, Week 4, Week 6, Week 8
Population: PD analysis population
Measure: Mean (Standard Deviation); unit: percent change in LDL-C
Arm/Group | Stayed at 5 mg: Tanner Stage 1 | Titrated to 10 mg: Tanner Stage 1 | Stayed at 10 mg: Tanner Stage 2+ | Titrated to 20 mg: Tanner Stage 2+
Number analyzed (Participants) | 5 | 10 | 9 | 15
percent change in LDL-C
  Week 2 | -36.27 (14.72) | -25.70 (7.76) | -38.14 (9.35) | -30.27 (9.22)
  Week 4 | -42.33 (8.24) | -30.27 (5.72) | -43.66 (7.78) | -35.13 (12.01)
  Week 6 | -38.87 (7.84) | -40.01 (6.34) | -41.22 (11.34) | -39.73 (10.40)
  Week 8 | -36.78 (11.16) | -42.70 (6.45) | -38.45 (7.84) | -40.39 (11.71)

4. Secondary Outcome: Absolute Change From Baseline in Total Cholesterol (TC)
Description: Total Cholesterol measured in millimoles per liter (mmol/L); assessments were performed in the fasting state (minimum 10-hour fast [optional at Weeks 2 and 6]). Change from baseline = value at observation minus baseline value.
Time Frame: Baseline, Week 2, Week 4, Week 6, Week 8
Population: PD analysis population
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Stayed at 5 mg: Tanner Stage 1 | Titrated to 10 mg: Tanner Stage 1 | Stayed at 10 mg: Tanner Stage 2+ | Titrated to 20 mg: Tanner Stage 2+
Number analyzed (Participants) | 5 | 10 | 9 | 15
mmol/L
  Baseline | 6.76 (0.46) | 8.58 (1.06) | 6.92 (0.71) | 8.40 (1.10)
  Week 2 | -1.89 (0.79) | -2.04 (0.69) | -2.11 (0.53) | -2.28 (0.82)
  Week 4 | -2.27 (0.63) | -2.24 (0.49) | -2.37 (0.61) | -2.66 (1.29)
  Week 6 | -2.03 (0.53) | -2.86 (0.79) | -2.28 (0.73) | -2.95 (1.19)
  Week 8 | -1.89 (0.44) | -3.20 (0.65) | -2.26 (0.69) | -3.22 (1.14)

5. Secondary Outcome: Percent Change From Baseline in Total Cholesterol (TC)
Description: Total cholesterol (TC): percent (%) change from baseline by treatment over time = [TC at observation minus TC at Week 0] divided by TC at Week 0 * 100. Assessments were performed in the fasting state (minimum 10-hour fast [optional at Weeks 2 and 6]).
Time Frame: Baseline, Week 2, Week 4, Week 6, Week 8
Population: PD analysis population
Measure: Mean (Standard Deviation); unit: percent change in TC
Arm/Group | Stayed at 5 mg: Tanner Stage 1 | Titrated to 10 mg: Tanner Stage 1 | Stayed at 10 mg: Tanner Stage 2+ | Titrated to 20 mg: Tanner Stage 2+
Number analyzed (Participants) | 5 | 10 | 9 | 15
percent change in TC
  Week 2 | -28.06 (11.23) | -24.11 (8.97) | -30.60 (7.49) | -26.78 (7.59)
  Week 4 | -33.37 (7.81) | -26.12 (4.24) | -33.98 (7.13) | -30.54 (11.60)
  Week 6 | -29.99 (8.00) | -33.12 (6.83) | -32.80 (8.97) | -34.06 (9.94)
  Week 8 | -27.80 (5.56) | -37.17 (5.28) | -32.43 (8.53) | -37.45 (9.89)

6. Secondary Outcome: Absolute Change From Baseline in Triglycerides (TG)
Description: Change from baseline in triglycerides measured in millimoles per liter (mmol/L); assessments were performed in the fasting state (minimum 10-hour fast [optional at Weeks 2 and 6]). Change from baseline = value at observation minus baseline value.
Time Frame: Baseline, Week 2, Week 4, Week 6, Week 8
Population: PD analysis population
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Stayed at 5 mg: Tanner Stage 1 | Titrated to 10 mg: Tanner Stage 1 | Stayed at 10 mg: Tanner Stage 2+ | Titrated to 20 mg: Tanner Stage 2+
Number analyzed (Participants) | 5 | 10 | 9 | 15
mmol/L
  Baseline | 0.76 (0.15) | 0.95 (0.27) | 1.03 (0.37) | 1.20 (0.50)
  Week 2 | 0.05 (0.34) | -0.08 (0.28) | 0.05 (0.68) | 0.00 (0.47)
  Week 4 | -0.05 (0.29) | -0.26 (0.30) | -0.10 (0.51) | -0.10 (0.37)
  Week 6 | 0.40 (0.62) | -0.04 (0.24) | -0.12 (0.42) | -0.04 (0.32)
  Week 8 | 0.02 (0.28) | -0.16 (0.37) | -0.31 (0.43) | -0.28 (0.41)

7. Secondary Outcome: Percent Change From Baseline in Triglycerides (TG)
Description: Triglycerides (TG): percent (%) change from baseline by treatment over time = [TG at observation minus TG at Week 0] divided by TG at Week 0 * 100. Assessments were performed in the fasting state (minimum 10-hour fast [optional at Weeks 2 and 6]).
Time Frame: Baseline, Week 2, Week 4, Week 6, Week 8
Population: PD analysis population
Measure: Mean (Standard Deviation); unit: percent change in TG
Arm/Group | Stayed at 5 mg: Tanner Stage 1 | Titrated to 10 mg: Tanner Stage 1 | Stayed at 10 mg: Tanner Stage 2+ | Titrated to 20 mg: Tanner Stage 2+
Number analyzed (Participants) | 5 | 10 | 9 | 15
percent change in TG
  Week 2 | 5.66 (38.26) | -6.87 (29.08) | 28.37 (85.32) | -0.56 (32.19)
  Week 4 | -6.20 (32.55) | -21.43 (30.42) | 1.27 (50.81) | -7.60 (25.75)
  Week 6 | 57.06 (78.73) | -1.27 (23.91) | -4.43 (32.52) | -2.72 (24.80)
  Week 8 | 1.69 (31.48) | -9.88 (33.31) | -20.94 (39.24) | -21.11 (23.85)

8. Secondary Outcome: Absolute Change From Baseline in High-Density Lipoprotein Cholesterol (HDL-C)
Description: Change from baseline in high-density lipoprotein cholesterol measured in millimoles per liter (mmol/L); assessments were performed in the fasting state (minimum 10-hour fast [optional at Weeks 2 and 6]). Change from baseline = value at observation minus baseline value.
Time Frame: Baseline, Week 2, Week 4, Week 6, Week 8
Population: PD analysis population
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Stayed at 5 mg: Tanner Stage 1 | Titrated to 10 mg: Tanner Stage 1 | Stayed at 10 mg: Tanner Stage 2+ | Titrated to 20 mg: Tanner Stage 2+
Number analyzed (Participants) | 5 | 10 | 9 | 15
mmol/L
  Baseline | 1.35 (0.12) | 1.45 (0.29) | 1.17 (0.18) | 1.18 (0.23)
  Week 2 | 0.08 (0.24) | -0.10 (0.29) | -0.05 (0.26) | -0.01 (0.20)
  Week 4 | -0.02 (0.05) | 0.00 (0.19) | 0.02 (0.21) | -0.01 (0.28)
  Week 6 | -0.12 (0.29) | -0.01 (0.18) | 0.04 (0.14) | -0.03 (0.23)
  Week 8 | 0.04 (0.22) | -0.07 (0.21) | 0.08 (0.25) | -0.08 (0.22)

9. Secondary Outcome: Percent Change From Baseline in High-Density Lipoprotein Cholesterol (HDL-C)
Description: High-density lipoprotein cholesterol (HDL-C): percent (%) change by treatment over time = [HDL-C at observation minus HDL-C at Week 0] divided by HDL-C at Week 0 * 100. Assessments were performed in the fasting state (minimum 10-hour fast [optional at Weeks 2 and 6]).
Time Frame: Baseline, Week 2, Week 4, Week 6, Week 8
Population: PD analysis population
Measure: Mean (Standard Deviation); unit: percent change in HDL-C
Arm/Group | Stayed at 5 mg: Tanner Stage 1 | Titrated to 10 mg: Tanner Stage 1 | Stayed at 10 mg: Tanner Stage 2+ | Titrated to 20 mg: Tanner Stage 2+
Number analyzed (Participants) | 5 | 10 | 9 | 15
percent change in HDL-C
  Week 2 | 5.38 (17.32) | -6.45 (21.01) | -4.11 (19.96) | -0.77 (17.66)
  Week 4 | -1.99 (3.90) | 1.59 (13.18) | 1.04 (17.38) | 1.77 (23.22)
  Week 6 | -10.18 (22.70) | -0.64 (10.35) | 3.28 (11.63) | -2.78 (21.49)
  Week 8 | 2.50 (15.02) | -2.84 (14.49) | 5.99 (21.02) | -5.19 (17.76)

10. Secondary Outcome: Absolute Change From Baseline in Apolipoprotein A-1 (Apo A-1)
Description: Change from baseline in Apolipoprotein A-1 measured in grams per liter (g/L); assessments were performed in the fasting state (minimum 10-hour fast [optional at Weeks 2 and 6]). Change from baseline = value at observation minus baseline value.
Time Frame: Baseline, Week 2, Week 4, Week 6, Week 8
Population: PD analysis population
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Stayed at 5 mg: Tanner Stage 1 | Titrated to 10 mg: Tanner Stage 1 | Stayed at 10 mg: Tanner Stage 2+ | Titrated to 20 mg: Tanner Stage 2+
Number analyzed (Participants) | 5 | 10 | 9 | 15
g/L
  Baseline | 1.42 (0.20) | 1.45 (0.20) | 1.29 (0.20) | 1.24 (0.15)
  Week 2 | 0.01 (0.17) | -0.08 (0.23) | -0.09 (0.22) | -0.01 (0.15)
  Week 4 | -0.09 (0.14) | -0.06 (0.13) | -0.06 (0.21) | 0.07 (0.29)
  Week 6 | -0.14 (0.18) | -0.02 (0.11) | -0.07 (0.19) | -0.04 (0.23)
  Week 8 | -0.03 (0.12) | -0.05 (0.13) | -0.04 (0.24) | -0.07 (0.21)

11. Secondary Outcome: Percent Change From Baseline in Apolipoprotein A-1 (Apo A-1)
Description: Apolipoprotein A-1 (Apo A-1): percent (%) change from baseline by treatment over time = [Apo A-1 at observation minus Apo A-1 at Week 0] divided by Apo A-1 at Week 0 * 100. Assessments were performed in the fasting state (minimum 10-hour fast [optional at Weeks 2 and 6]).
Time Frame: Baseline, Week 2, Week 4, Week 6, Week 8
Population: PD analysis population
Measure: Mean (Standard Deviation); unit: percent change in Apo A-1
Arm/Group | Stayed at 5 mg: Tanner Stage 1 | Titrated to 10 mg: Tanner Stage 1 | Stayed at 10 mg: Tanner Stage 2+ | Titrated to 20 mg: Tanner Stage 2+
Number analyzed (Participants) | 5 | 10 | 9 | 15
percent change in Apo A-1
  Week 2 | 1.69 (11.21) | -5.24 (15.86) | -5.96 (16.76) | -0.53 (11.90)
  Week 4 | -5.15 (8.20) | -3.30 (8.11) | -3.73 (16.43) | 7.54 (25.24)
  Week 6 | -9.90 (14.01) | -0.97 (7.04) | -4.21 (14.81) | -2.82 (18.20)
  Week 8 | -1.24 (8.49) | -3.37 (9.35) | -2.60 (20.22) | -4.82 (16.13)

12. Secondary Outcome: Absolute Change From Baseline in Apolipoprotein B (Apo B)
Description: Change from baseline in Apolipoprotein B measured in grams per liter (g/L); assessments were performed in the fasting state (minimum 10-hour fast [optional at Weeks 2 and 6]). Change from baseline = value at observation minus baseline value.
Time Frame: Baseline, Week 2, Week 4, Week 6, Week 8
Population: PD analysis population
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Stayed at 5 mg: Tanner Stage 1 | Titrated to 10 mg: Tanner Stage 1 | Stayed at 10 mg: Tanner Stage 2+ | Titrated to 20 mg: Tanner Stage 2+
Number analyzed (Participants) | 5 | 10 | 9 | 15
g/L
  Baseline | 1.09 (0.13) | 1.49 (0.24) | 1.26 (0.14) | 1.52 (0.18)
  Week 2 | -0.23 (0.13) | -0.31 (0.19) | -0.39 (0.14) | -0.42 (0.16)
  Week 4 | -0.33 (0.11) | -0.40 (0.13) | -0.44 (0.10) | -0.47 (0.22)
  Week 6 | -0.27 (0.15) | -0.53 (0.17) | -0.42 (0.15) | -0.52 (0.18)
  Week 8 | -0.30 (0.08) | -0.59 (0.15) | -0.41 (0.17) | -0.49 (0.30)

13. Secondary Outcome: Percent Change From Baseline in Apolipoprotein B (Apo B)
Description: Apolipoprotein B (Apo B): percent (%) change from baseline by treatment over time = [Apo B at observation minus Apo B at Week 0] divided by Apo B at Week 0 * 100. Assessments were performed in the fasting state (minimum 10-hour fast [optional at Weeks 2 and 6]).
Time Frame: Baseline, Week 2, Week 4, Week 6, Week 8
Population: PD analysis population
Measure: Mean (Standard Deviation); unit: percent change in Apo B
Arm/Group | Stayed at 5 mg: Tanner Stage 1 | Titrated to 10 mg: Tanner Stage 1 | Stayed at 10 mg: Tanner Stage 2+ | Titrated to 20 mg: Tanner Stage 2+
Number analyzed (Participants) | 5 | 10 | 9 | 15
percent change in Apo B
  Week 2 | -21.92 (13.97) | -19.88 (10.96) | -30.81 (10.27) | -27.46 (8.89)
  Week 4 | -29.89 (8.94) | -26.56 (5.33) | -34.69 (6.10) | -30.42 (11.86)
  Week 6 | -24.58 (12.96) | -35.26 (6.85) | -33.26 (10.38) | -33.61 (9.59)
  Week 8 | -27.39 (5.97) | -39.59 (5.83) | -31.94 (11.64) | -31.26 (18.57)

14. Secondary Outcome: Absolute Change From Baseline in Very Low-density Lipoprotein-cholesterol (VLDL-C)
Description: Change from baseline in very low-density lipoprotein-cholesterol (VLDL-C) measured in millimoles per liter (mmol/L). Change from baseline = value at observation minus baseline value. Assessments were performed in the fasting state (minimum 10-hour fast [optional at Weeks 2 and 6]).
Time Frame: Baseline, Week 2, Week 4, Week 6, Week 8
Population: PD analysis population
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Stayed at 5 mg: Tanner Stage 1 | Titrated to 10 mg: Tanner Stage 1 | Stayed at 10 mg: Tanner Stage 2+ | Titrated to 20 mg: Tanner Stage 2+
Number analyzed (Participants) | 5 | 10 | 9 | 15
mmol/L
  Baseline | 0.54 (0.15) | 0.76 (0.30) | 0.65 (0.11) | 0.99 (0.31)
  Week 2 | -0.22 (0.12) | -0.31 (0.38) | -0.12 (0.29) | -0.38 (0.33)
  Week 4 | -0.18 (0.24) | -0.30 (0.27) | -0.14 (0.24) | -0.39 (0.35)
  Week 6 | -0.01 (0.17) | -0.28 (0.32) | -0.20 (0.17) | -0.36 (0.28)
  Week 8 | -0.13 (0.32) | -0.42 (0.28) | -0.35 (0.14) | -0.55 (0.32)

15. Secondary Outcome: Percent Change From Baseline in Very Low-density Lipoprotein-cholesterol (VLDL-C)
Description: Very low-density lipoprotein-cholesterol (VLDL-C): percent (%) change from baseline by treatment over time = [VLDL-C at observation minus VLDL-C at Week 0] divided by VLDL-C at Week 0 * 100. Assessments were performed in the fasting state (minimum 10-hour fast [optional at Weeks 2 and 6]).
Time Frame: Baseline, Week 2, Week 4, Week 6, Week 8
Population: PD analysis population
Measure: Mean (Standard Deviation); unit: percent change in VLDL-C
Arm/Group | Stayed at 5 mg: Tanner Stage 1 | Titrated to 10 mg: Tanner Stage 1 | Stayed at 10 mg: Tanner Stage 2+ | Titrated to 20 mg: Tanner Stage 2+
Number analyzed (Participants) | 5 | 10 | 9 | 15
percent change in VLDL-C
  Week 2 | -42.20 (25.17) | -28.49 (43.50) | -14.50 (41.19) | -39.95 (37.24)
  Week 4 | -30.66 (48.66) | -31.86 (37.62) | -21.10 (37.56) | -36.35 (28.79)
  Week 6 | 4.10 (36.46) | -25.59 (44.90) | -29.20 (25.11) | -35.08 (25.06)
  Week 8 | -12.31 (57.38) | -50.29 (21.44) | -53.61 (19.21) | -52.38 (29.34)

16. Secondary Outcome: Absolute Change From Baseline in Flow-Mediated Dilatation at Week 8
Description: Brachial artery flow-mediated dilatation (FMD) = (max minus baseline diameter divided by baseline diameter) x 100%. Standardized image acquisition: brachial artery images recorded for one minute at rest, blood pressure cuff inflated to 250 mm Hg for 5 minutes with brachial artery imaged continuously throughout cuff inflation, cuff released to produce reactive hyperaemia and the brachial artery imaged continuously for 3 minutes after release. Total duration of measurement approximately 25 minutes. Change from baseline = value at observation minus baseline value.
Time Frame: Baseline, Week 8
Population: PD analysis population. Flow-mediated dilation (FMD) was measured at centers with established FMD facilities.
Measure: Mean (Standard Deviation); unit: FMD
Arm/Group | Stayed at 5 mg: Tanner Stage 1 | Titrated to 10 mg: Tanner Stage 1 | Stayed at 10 mg: Tanner Stage 2+ | Titrated to 20 mg: Tanner Stage 2+
Number analyzed (Participants) | 4 | 7 | 5 | 12
FMD
  Baseline | 4.34 (3.15) | 7.41 (3.30) | 5.05 (3.86) | 3.67 (2.51)
  Week 8 | -0.16 (2.32) | -1.14 (1.47) | -0.32 (4.83) | 1.35 (2.73)

17. Secondary Outcome: Percent Change From Baseline in Flow-Mediated Dilatation at Week 8
Description: Brachial Flow-Mediated Dilatation (FMD) = (max minus baseline diameter divided by baseline diameter) x 100%.
  .
Time Frame: Baseline, Week 8
Population: PD analysis population. Flow-mediated dilation (FMD) was measured at centers with established FMD facilities.
Measure: Mean (Standard Deviation); unit: percent change in FMD
Arm/Group | Stayed at 5 mg: Tanner Stage 1 | Titrated to 10 mg: Tanner Stage 1 | Stayed at 10 mg: Tanner Stage 2+ | Titrated to 20 mg: Tanner Stage 2+
Number analyzed (Participants) | 4 | 7 | 5 | 12
percent change in FMD | -17.19 (23.67) | -20.77 (37.03) | -9.77 (63.20) | 1.49 (28.64)

18. Primary Outcome: Parent-metabolite Population Pharmacokinetic (PK) Model for Atorvastatin and Its Metabolites: Apparent Volume of Distribution of the Central Compartment (Vc/F)
Description: Parent-metabolite population PK model built using sparse blood samples from Tanner Stages 1 and 2+. Sampling times: Weeks 2 + 6: single sample between 4 -12 hours postdose; Weeks 4 + 8: predose, 1 + 2 hours postdose. Plasma samples analyzed for atorvastatin and active hydroxyacid metabolite (o-hydroxyatorvastatin) concentrations using validated, sensitive, specific high-performance liquid chromatography tandem mass spectrometric method. Vc/F value based on 70 kg body weight. Parameter estimation uncertainty (95% CI) by non-parametric bootstrap analysis. Data presented are result of model used.
Time Frame: Week 2, Week 4, Week 6, Week 8
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: liters
Groups:
- Atorvastatin (5 mg, 10 mg, 20 mg): Tanner Stages 1 and 2+: Tanner Stage 1: Initial dose 5 mg/day through Week 4; after Week 4 dose may have been doubled to 10 mg/day if target LDL-C was not attained and study drug was well tolerated; Tanner Stage 2+: Initial dose 10 mg/day through Week 4; after Week 4 dose may have been doubled to 20 mg/day if target LDL-C was not attained and study drug was well tolerated.
Arm/Group | Atorvastatin (5 mg, 10 mg, 20 mg): Tanner Stages 1 and 2+
Number analyzed (Participants) | 39
liters | 1020 [209 to 2210]

ADVERSE EVENTS:
Groups:
- All Subjects (5 mg, 10 mg): Tanner Stage 1: Atorvastatin: subjects who stayed at initial dose of 5 mg/day for duration of study and subjects who titrated after Week 4 to 10 mg/day if target LDL-C was not attained and study drug was well tolerated.
- All Subjects (10 mg, 20 mg): Tanner Stage 2+: Atorvastatin: subjects who stayed at initial dose of 10 mg/day for duration of study and subjects who titrated to 20 mg/day after Week 4 if target LDL-C was not attained and study drug was well tolerated.
Arm/Group | All Subjects (5 mg, 10 mg): Tanner Stage 1 | All Subjects (10 mg, 20 mg): Tanner Stage 2+
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/24
Other Adverse Events (participants affected / at risk) | 9/15 | 13/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Subjects (5 mg, 10 mg): Tanner Stage 1 (N=15) | All Subjects (10 mg, 20 mg): Tanner Stage 2+ (N=24)
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0
Pain (General disorders) | 0 | 1
Bronchopneumonia (Infections and infestations) | 1 | 0
Ear infection (Infections and infestations) | 0 | 1
Gastritis viral (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 1
Influenza (Infections and infestations) | 0 | 1
Lower respiratory tract infection bacterial (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 1 | 2
Tonsillitis (Infections and infestations) | 0 | 1
Viral rhinitis (Infections and infestations) | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 3 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 2
Blood creatinine increased (Investigations) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Headache (Nervous system disorders) | 2 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of < 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), < 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.